CLINICAL TRIAL: NCT00141388
Title: Pregabalin Open-Label Add-On Trial: An Open-Label, Multicenter Follow-On Study to Determine Long-Term Safety and Efficacy in Patients With Partial Seizures.
Brief Title: To Evaluate the Long-Term Safety and Efficacy of Pregabalin in Patients With Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-010
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Seizure Disorder, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate the long-term safety and efficacy of pregabalin in patients with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for the preceding double-blind study
* Have received double-blind study medication and wish to receive open-label pregabalin.

Exclusion Criteria:

* Cannot have absence seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 1998-07; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (43):
- United States (36):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Spring Hill, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Greenbelt, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Bennington, Vermont
- Canada (7):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Edmont, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec